CLINICAL TRIAL: NCT01664923
Title: STRIVE: A MULTICENTER PHASE 2, RANDOMIZED, DOUBLE-BLIND, EFFICACY AND SAFETY STUDY OF ENZALUTAMIDE VS. BICALUTAMIDE IN MEN WITH PROSTATE CANCER WHO HAVE FAILED PRIMARY ANDROGEN DEPRIVATION THERAPY
Brief Title: Safety and Efficacy Study of Enzalutamide Versus Bicalutamide in Men With Prostate Cancer
Acronym: STRIVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Astellas Pharma Inc (Industry); Medivation LLC, a wholly owned subsidiary of Pfizer Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MDV3100-09; C3431014 (Other: Alias Study Number)
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; enzalutamide; MDV3100
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; bicalutamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Enzalutamide (Experimental): Enzalutamide 160 mg/day orally
  Interventions: Drug: Enzalutamide
- Bicalutamide (Active Comparator): 50 mg/day orally
  Interventions: Drug: Bicalutamide

INTERVENTIONS:
Drug: Enzalutamide — 160 mg, daily, by mouth.
  Other Names: MDV3100; Xtandi
  Arms: Enzalutamide
Drug: Bicalutamide — 50 mg, daily, by mouth
  Other Names: Casodex
  Arms: Bicalutamide

SUMMARY:
The purpose of this study is to determine the safety and efficacy of enzalutamide vs bicalutamide in asymptomatic or mildly symptomatic patients with prostate cancer who have disease progression despite primary androgen deprivation therapy.

DETAILED DESCRIPTION:
This study is a multicenter phase 2, randomized, double-blind, efficacy and safety study of enzalutamide (160 mg/day) vs. bicalutamide (50 mg/day) in patients with recurrent prostate cancer who have serologic and/or radiographic disease progression despite primary androgen deprivation therapy.

Throughout the study, safety and tolerability will be assessed by the recording of adverse events, monitoring of vital signs, physical examinations, and safety laboratory evaluations.

Following study unblinding, study patients receiving enzalutamide or bicalutamide at the time of unblinding and qualifying patients randomized to bicalutamide who discontinued prior to unblinding will be offered the opportunity to receive open label enzalutamide treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males age 18 or older;
* Histologically or cytologically confirmed adenocarcinoma of the prostate;
* Ongoing androgen deprivation therapy;
* Serum testosterone level ≤ 50 ng/dL (1.73 nmol/L) at the Screening visit;
* Progressive disease at study entry defined by prostate-specific antigen (PSA) progression and/or radiographic progression that occurred while the patient was on primary androgen deprivation therapy;
* Asymptomatic or mildly symptomatic from prostate cancer;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
* Estimated life expectancy of ≥ 12 months;
* Able to swallow the study drug and comply with study requirements.

Exclusion Criteria:

* Severe concurrent disease, infection, or co-morbidity;
* Known or suspected brain metastasis or active leptomeningeal disease;
* History of another invasive malignancy within the previous 5 years other than treated non-melanomatous skin cancer and American Joint Committee on Cancer (AJCC) Stage 0 or Stage 1 cancers that have a remote probability of recurrence;
* Absolute neutrophil count < 1,500/µL, or platelet count < 100,000/µL, or hemoglobin < 9 g/dL at the Screening visit;
* Total bilirubin, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 times the upper limit of normal (ULN) at the Screening visit;
* Creatinine > 2 mg/dL at the Screening visit;
* Albumin < 3.0 g/dL at the Screening visit;
* History of seizure or any condition that may predispose to seizure;
* Clinically significant cardiovascular disease;
* Gastrointestinal disorder affecting absorption (e.g., gastrectomy, active peptic ulcer disease within last 3 months);
* Major surgery within 4 weeks of enrollment;
* Use of opiate analgesics for pain from prostate cancer within 4 weeks of enrollment;
* Radiation therapy for treatment of the primary tumor within 3 weeks of enrollment;
* Prior radiation or radionuclide therapy for treatment of distant metastases;
* Prior ketoconazole, abiraterone, or cytotoxic chemotherapy for prostate cancer;
* Treatment with hormonal therapy or biologic therapy for prostate cancer within 4 weeks of enrollment;
* Use of antiandrogens within 4 weeks prior to enrollment;
* Prior disease progression, as assessed by the Investigator, while receiving bicalutamide;
* Participation in a previous clinical trial of enzalutamide or an investigational agent that inhibits the androgen receptor or androgen synthesis (patients who received placebo are acceptable);
* Use of an investigational agent within 4 weeks of enrollment;
* Use of herbal products that may have hormonal anti-prostate cancer activity and/or are known to decrease PSA levels (e.g., saw palmetto) or systemic corticosteroids for prostate cancer within 4 weeks of enrollment;
* Any condition or reason that, in the opinion of the Investigator, interferes with the ability of the patient to participate in the trial, which places the patient at undue risk, or complicates the interpretation of safety data.

Open-Label Treatment Period:

Inclusion Criteria:

* Received randomized double blind treatment in MDV3100-09 as follows:

  * Randomized to enzalutamide and receiving enzalutamide at the time of study unblinding;
  * Randomized to bicalutamide and receiving bicalutamide at the time of study unblinding;
  * Randomized to bicalutamide and discontinued bicalutamide before study unblinding;
* Willing to maintain androgen deprivation therapy with a gonadotropin releasing hormone (GnRH) agonist/antagonist or has had a bilateral orchiectomy.

Exclusion Criteria:

* Is currently or has taken commercially available enzalutamide (Xtandi) prior to participation in this open-label extension;
* Discontinued enzalutamide during the double-blind portion of the study prior to unblinding;
* Has any clinically significant cardiovascular, dermatologic, endocrine, gastrointestinal, hematologic, hepatic, infectious, metabolic, neurologic, psychiatric, psychologic, pulmonary, or renal disorder or any other condition, including excessive alcohol or drug abuse, or secondary malignancy, that may interfere with study participation in the opinion of the investigator or medical monitor;
* Has a current or previously treated brain metastasis or leptomeningeal disease;
* Has a history of seizure or any condition that may predispose to seizure (eg, prior cortical stroke or significant brain trauma);
* Has a history of loss of consciousness or transient ischemic attack within 12 months of open label day 1;
* Has taken cytotoxic chemotherapy or investigational therapy within 4 weeks before enrollment (open label day 1).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 396 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (104):
- United States (104):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Alabama at Birmingham，IDS Pharmacy, Birmingham, Alabama
  - Desert Springs Cancer Care, Scottsdale, Arizona
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - Urological Associates of Southern Arizona, PC, Tucson, Arizona
  - Southern California Permanente Medical Group, Anaheim, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Antioch, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Fairfield, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Gilroy, California
  - Southern California Permanente Medical Group, Los Angeles, California
  - Tower Urology, Los Angeles, California
  - UCLA Clark Urology Clinic, Los Angeles, California
  - UCLA Department of Pharmaceutical Services, Los Angeles, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Martinez, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Milpitas, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Modesto, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Moutain View, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Napa, California
  - Kaiser Permanente Medical Center, Oakland, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Pleasanton, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Redwood City, California
  - Kaiser Permanente Medical Center, Roseville, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - UC Davis Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center, Sacramento, California
  - San Bernardino Urological Associates Medical Group, San Bernardino, California
  - Southern California Permanente Medical Group, San Diego, California
  - Kaiser Permanente Medical Center, San Francisco, California
  - Kaiser Permanente Medical Center, San Jose, California
  - Kaiser Permanente Medical Center, San Leandro, California
  - Southern California Permanente Medical Group, San Marcos, California
  - Kaiser Permanente Medical Center, Santa Clara, California
  - Skyline Urology, Sherman Oaks, California
  - Kaiser Permanente Medical Center, South San Francisco, California
  - Standford Health Care, Stanford, California
  - Skyline Urology, Torrance, California
  - Kaiser Permanente Medical Center, Vallejo, California
  - Kaiser Permanente Medical Center, Walnut Creek, California
  - Anschutz Cancer Center Pavilion Pharmacy, Aurora, Colorado
  - Anschutz Inpatient Pavilion, Aurora, Colorado
  - University of Colorado Cancer Center, Anschutz Cancer Pavilion, Aurora, Colorado
  - The Urology Center of Colorado, Denver, Colorado
  - George Washington University - Medical Faculty Associates, Washington D.C., District of Columbia
  - Advanced Urology institute, Daytona Beach, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - Specialists In Urology, Naples, Florida
  - First Urology, PSC, Jeffersonville, Indiana
  - Metairie Oncologist, LLC, Metairie, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Regional Urology, LLC, Shreveport, Louisiana
  - Chesapeake Urology Research Associates, Towson, Maryland
  - Michigan Institute of Urology, Troy, Michigan
  - Minnesota Oncology Hematology, P.A., Edina, Minnesota
  - Minnesota Oncology Hematology, P.A., Woodbury, Minnesota
  - Barnes-Jewish West County Hospital, Creve Coeur, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University Infusion Center Pharmacy, St Louis, Missouri
  - Washington University, School of Medicine, 7th Floor, Center for Advanced Medicine, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - GU Research network,LLC / Urology Cancer Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - AccuMed Research Associates, Garden City, New York
  - Premier Medical Group of the Hudson Valley PC, Poughkeepsie, New York
  - Associated Medical Professionals of NY, PLLC, Syracuse, New York
  - Carolinas Medical Center-Steelcreek, Charlotte, North Carolina
  - Carolina Clinical Trials, LLC, Concord, North Carolina
  - Carolina Urology Partners, PLLC, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Investigational Chemotherapy Services, Durham, North Carolina
  - Alliance Urology Specialists, PA, Greensboro, North Carolina
  - Rowan Regional Medical Center, Salisbury, North Carolina
  - Wake Forest Baptist Health Urology, Winston-Salem, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - TriState Urologic Services PSC Inc., dba The Urology Group, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Cleveland, Ohio
  - Peace Harbor Hospital, Florence, Oregon
  - Salem Hospital, Salem, Oregon
  - Oregon Urology Institute, Springfield, Oregon
  - Sacred Heart Nuclear Medicine, Springfield, Oregon
  - Lancaster Urology, Lancaster, Pennsylvania
  - Jefferson Medical Oncology, Philadelphia, Pennsylvania
  - Jefferson Urology Associates, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC Cancer Center Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Mount Nittany Physician Group, State College, Pennsylvania
  - Mount Nittany Health, State College, Pennsylvania
  - Charleston Hematology Oncology Associates, PA, Charleston, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Associates P.C., Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Urology Clinics of North Texas, Dallas, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology-Memorial City, Houston, Texas
  - Urology San Antonio Research, San Antonio, Texas
  - University of Utah/Huntsman Cancer Hospital, Salt Lake City, Utah
  - University of Utah/Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Oncology Associates, Hampton, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Urology of Virginia, PLLC., Virginia Beach, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Clinical Sciences Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Penson DF, Armstrong AJ, Concepcion RS, Agarwal N, Olsson CA, Karsh LI, Dunshee CJ, Duggan W, Shen Q, Sugg J, Haas GP, Higano CS. Enzalutamide versus bicalutamide in patients with nonmetastatic castration-resistant prostate cancer: a prespecified subgroup analysis of the STRIVE trial. Prostate Cancer Prostatic Dis. 2022 Feb;25(2):363-365. doi: 10.1038/s41391-021-00465-7. Epub 2021 Oct 7. PMID 34621011
- [Derived] Schultz NM, Shore ND, Chowdhury S, Klotz LH, Concepcion RS, Penson DF, Karsh LI, Yang H, Brown BA, Barlev A, Flanders SC. Number-needed-to-treat analysis of clinical progression in patients with metastatic castration-resistant prostate cancer in the STRIVE and TERRAIN trials. BMC Urol. 2018 Sep 6;18(1):77. doi: 10.1186/s12894-018-0387-7. PMID 30189902
- [Derived] Penson DF, Armstrong AJ, Concepcion R, Agarwal N, Olsson C, Karsh L, Dunshee C, Wang F, Wu K, Krivoshik A, Phung D, Higano CS. Enzalutamide Versus Bicalutamide in Castration-Resistant Prostate Cancer: The STRIVE Trial. J Clin Oncol. 2016 Jun 20;34(18):2098-106. doi: 10.1200/JCO.2015.64.9285. Epub 2016 Jan 25. PMID 26811535

RESULTS

PARTICIPANT FLOW:
Groups:
- Enzalutamide: Participants received enzalutamide 160 milligram (mg), self-administered as four 40-mg capsules, and 1 bicalutamide matching placebo capsule once per day, by mouth for up to 29 months in double blind (DB) phase. Participants who completed DB phase and consented to participate in open label phase, received enzalutamide 160 mg, self-administered as four 40-mg capsules once per day by mouth for up to 36 months in open label phase.
- Bicalutamide Then Enzalutamide: Participants received bicalutamide 50 mg, self-administered as 1 capsule, once per day by mouth and 4 enzalutamide matching placebo capsules for up to 29 months in DB phase. Participants who completed DB phase and consented to participate in open label phase, received enzalutamide 160 mg, self-administered as four 40-mg capsules, once per day by mouth for up to 36 months in open label phase.
Period: Period1:Double Blind Phase-29 Months
Arm/Group | Enzalutamide | Bicalutamide Then Enzalutamide
Started | 198 | 198
Received Study Treatment | 197 | 198
Completed | 93 | 38
Not Completed | 105 | 160
Not completed — Death | 8 | 6
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 12 | 8
Not completed — Disease Progression | 65 | 132
Not completed — Adverse Event | 14 | 9
Not completed — Other | 3 | 4
Not completed — Randomized, But Not treated | 1 | 0
Period: Period 2: Open-label Phase-36 Months
Arm/Group | Enzalutamide | Bicalutamide Then Enzalutamide
Started | 93 | 38
Treated | 93 | 37
Completed | 52 | 15
Not Completed | 41 | 23
Not completed — Death | 3 | 1
Not completed — On Treatment | 1 | 1
Not completed — Disease progression | 28 | 9
Not completed — Other | 3 | 1
Not completed — Adverse Event | 4 | 7
Not completed — Withdrawal by Subject | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Enzalutamide: Participants received enzalutamide 160 mg, self-administered as four 40-mg capsules, once per day by mouth and 1 bicalutamide-placebo capsule in DB phase.
- Bicalutamide: Participants received bicalutamide 50 mg, self-administered as 1 capsule, once per day by mouth and 4 enzalutamide-placebo capsules in DB phase.
- Total: Total of all reporting groups
Arm/Group | Enzalutamide | Bicalutamide | Total
Number analyzed (Participants) | 198 | 198 | 396
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 39 | 25 | 64
  65-74 years | 82 | 76 | 158
  ≥ 75 years | 77 | 97 | 174
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 198 | 198 | 396
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 198 | 198 | 396

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as time from randomization to earliest objective evidence of prostate specific-antigen (PSA) progression, radiographic progression, or death on study. PSA progression was defined as ≥ 25% increase in PSA with an absolute increase ≥ 2 ng/mL above the nadir and was to be confirmed by a second consecutive assessment. Radiographic progression in bone was based on The Prostate Cancer Clinical Trials Working Group (PCWG2) guidelines defined as at least 2 new lesions on bone scan. Radiographic progression in soft tissue on Computerized Tomography/Magnetic Resonance Imaging (CT/MRI) was based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). CT/MRI and bone scans were read locally by the same radiologist (or nuclear medicine physician for interpretation of bone scans) whenever possible. Participants not known to have had a PFS event at the time of the analysis data cutoff were censored at the date of last assessment.
Time Frame: From randomization until the data cut-off date of 09 February 2015, median duration of treatment was 14.7 months in the enzalutamide arm and 8.4 months in the bicalutamide arm.
Population: Intent-to-treat population: all participants randomly assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide | Bicalutamide
Number analyzed (Participants) | 198 | 198
months | 19.4 [16.5 to NA] — The upper limit of the 95% confidence interval was not available because an insufficient number of participants had an event at the time of analysis. | 5.7 [5.6 to 8.1]
Statistical Analysis 1: Comparison: Enzalutamide vs Bicalutamide; Test type: Superiority or Other; p < 0.0001, Log Rank — P-value based on log-rank test stratified by disease stage at study entry as reported on the case report form (CRF); Hazard Ratio (HR) = 0.240, 95% CI 2-sided [0.181 to 0.320] — Hazard ratio is based on a Cox regression model (with treatment as the only covariate) stratified by disease stage at study entry and is relative to bicalutamide with < 1 favoring enzalutamide

2. Secondary Outcome: Time to PSA Progression
Description: PSA progression was defined as ≥ 25% increase in PSA with an absolute increase ≥ 2 ng/mL above the nadir and was to be confirmed by a second consecutive assessment at least 3 weeks later. Participants not known to have had PSA progression were censored at the date of last PSA assessment.
Time Frame: as for outcome 1
Population: Intent-to-treat population: all participants randomly assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide | Bicalutamide
Number analyzed (Participants) | 198 | 198
months | NA [19.4 to NA] — The median time to PSA progression and its upper limit of the 95% confidence interval were not available because an insufficient number of participants had an event at the time of analysis. | 8.3 [5.7 to 8.5]
Statistical Analysis 1: Comparison: Enzalutamide vs Bicalutamide; Test type: Superiority or Other; p < 0.0001, Log Rank — P-value based on log-rank test stratified by disease stage at study entry as reported on the CRF; Hazard Ratio (HR) = 0.190, 95% CI 2-sided [0.137 to 0.264] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants With a PSA Response ≥ 50%
Description: PSA response was defined as a reduction in PSA of at least 50% from baseline at any post baseline assessment confirmed by a second PSA assessment at least 3 weeks later.
Time Frame: as for outcome 1
Population: Evaluable intent-to-treat population: all participants randomly assigned to study treatment and had a baseline and at least 1 post baseline PSA measurement.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzalutamide | Bicalutamide
Number analyzed (Participants) | 192 | 195
percentage of participants | 81.3 [75.0 to 86.5] | 31.3 [24.8 to 38.3]
Statistical Analysis 1: Comparison: Enzalutamide vs Bicalutamide; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Comparison of the 2 treatment groups using the Cochran-Mantel-Haenszel mean score test stratified by disease stage at study entry; Difference in rates = 50.0, 95% CI 2-sided [41.4 to 58.5] — Enzalutamide response rate minus bicalutamide response rate

4. Secondary Outcome: Duration of Radiographic PFS
Description: Duration of radiographic PFS was defined as the time from randomization to the earliest objective evidence of radiographic disease progression or death on study and was to be evaluated for participants with metastatic disease at study entry. Radiographic disease progression in bone was based on PCWG2 guidelines defined as at least 2 new lesions on bone scan. Radiographic disease progression in soft tissue on CT/MRI was based on RECIST 1.1. CT/MRI and bone scans were read locally by the same radiologist (or nuclear medicine physician for interpretation of bone scans) whenever possible. Participants not known to have had radiographic progression at the time of analysis data cutoff were censored at the date of last radiographic assessment.
Time Frame: as for outcome 1
Population: All participants with metastatic disease at study entry and randomly assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide | Bicalutamide
Number analyzed (Participants) | 128 | 129
months | NA [16.7 to NA] — The median duration of radiographic PFS and its upper limit of the 95% confidence interval were not available because an insufficient number of participants had an event at the time of analysis. | 8.3 [8.1 to 11.1]
Statistical Analysis 1: Comparison: Enzalutamide vs Bicalutamide; Test type: Superiority or Other; p < 0.0001, Log Rank; P-value is based on an unstratified log-rank test; Hazard Ratio (HR) = 0.324, 95% CI 2-sided [0.211 to 0.497] — Hazard ratio is based on an unstratified Cox-regression model (with treatment as the only covariate) and is relative to bicalutamide with < 1 favoring enzalutamide

5. Secondary Outcome: Quality of Life: Time to Degradation of Functional Assessment of Cancer Therapy - Prostate (FACT-P)
Description: The FACT-P is a multidimensional, self-reported quality of life instrument consisting of 27 core items that assess patient function in 4 domains: physical, social/family, emotional, and functional well-being, and supplemented by 12 site-specific items to assess for prostate-related symptoms. Each item is rated on a 0 to 4 Likert-type scale, and then combined to produce subscale scores for each domain, as well as a global quality of life score (0 to 156) with higher scores representing better quality of life. Time to degradation of FACT-P was defined as the time from randomization to first assessment with at least a 10-point decrease from baseline in the global FACT-P score for each participant. Participants with no score degradation at the time of analysis data cutoff were censored at the date of last assessment showing no degradation.
Time Frame: as for outcome 1
Population: Intent-to-treat population: all participants randomly assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide | Bicalutamide
Number analyzed (Participants) | 198 | 198
months | 8.4 [6.3 to 11.4] | 8.3 [6.1 to 11.1]
Statistical Analysis 1: Comparison: Enzalutamide vs Bicalutamide; Test type: Superiority or Other; p = 0.4945, Log Rank — This secondary endpoint was not adjusted for multiple comparisons; P-value is based on a log-rank test stratified by disease stage at study entry; Hazard Ratio (HR) = 0.910, 95% CI 2-sided [0.695 to 1.192] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Best Overall Soft Tissue Response
Description: Best overall soft tissue response is defined as partial response (PR) or complete response (CR) while on study treatment based on investigator assessment of target, nontarget, and new lesions using RECIST 1.1. Only participants in the metastatic population with measurable soft tissue disease (at least 1 target lesion identified per RECIST 1.1) at screening were included in the analysis. All percentages are based on number of participants with metastatic and measurable soft tissue disease at screening in each treatment group.
Time Frame: as for outcome 1
Population: All participants who were randomly assigned to study treatment and had metastatic and measurable soft tissue disease at screening.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzalutamide | Bicalutamide
Number analyzed (Participants) | 35 | 43
percentage of participants | 60.0 [42.11 to 76.13] | 14.0 [5.30 to 27.93]
Statistical Analysis 1: Comparison: Enzalutamide vs Bicalutamide; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — This secondary endpoint was not adjusted for multiple comparisons; Based on unstratified Cochran-Mantel-Haenszel mean score test; Difference in objective response rate = 46.05, 95% CI 2-sided [26.79 to 65.30]

7. Secondary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. An SAE was an AE resulting in any of following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), persistent or significant disability or incapacity, congenital anomaly. A treatment emergent AE defined as an event that emerged during treatment period (From first dose of study drug until end of open label phase [up to maximum duration of 65 months]) that was absent before treatment, or worsened during treatment period relative to pre-treatment state. AE included both serious and non- SAE. Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An AE was considered related to study drug if event was assessed by investigator as probably or possibly related.
Time Frame: From first dose of study drug until the end of open label phase (up to maximum duration of 65 months)
Population: Safety population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Enzalutamide: Participants received enzalutamide 160 mg, self-administered as four 40-mg capsules, and 1 bicalutamide matching placebo capsule once per day, by mouth for up to 29 months in DB phase. Participants who completed DB phase and consented to participate in open label phase, received enzalutamide 160 mg, self-administered as four 40-mg capsules once per day by mouth for up to 36 months in open label phase.
- DB Phase: Bicalutamide: Participants received bicalutamide 50 mg, self-administered as 1 capsule, once per day by mouth and 4 enzalutamide matching placebo capsules for up to 29 months in DB phase.
- Open Label Phase: Bicalutamide Crossover to Enzalutamide: Participants who received bicalutamide 50 mg in DB phase and consented to participate in open label phase, received enzalutamide 160 mg, self-administered as four 40-mg capsules, once per day by mouth in open label phase for up to 36 months.
Arm/Group | Enzalutamide | DB Phase: Bicalutamide | Open Label Phase: Bicalutamide Crossover to Enzalutamide
Number analyzed (Participants) | 197 | 198 | 37
percentage of participants
  Any AE | 96.4 | 90.4 | 97.3
  AE Leading to Study Drug Discontinuation | 16.2 | 13.1 | 24.3
  AE Leading to Death | 4.6 | 3.0 | 8.1
  Serious AE | 38.6 | 30.3 | 43.2
  AE Related to Study Drug | 66.5 | 53.5 | 70.3
  Serious AE Related to Study Drug | 7.6 | 3.5 | 2.7

ADVERSE EVENTS:
Time Frame: From first dose of study drug until the end of open label phase (up to maximum duration of 65 months)
Description: Same event may appear as AE and SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study
Groups:
- Enzalutamide: Participants received enzalutamide 160 mg, self-administered as four 40-mg capsules, once per day by mouth and 1 bicalutamide-placebo capsule for up to 29 months in DB phase. Participants who completed DB phase and consented to participate in open label phase, received same treatment for up to 36 months in open label phase.
- DB Phase: Bicalutamide: Participants received bicalutamide 50 mg, self-administered as 1 capsule, once per day by mouth and 4 enzalutamide-placebo capsules for up to 29 months in DB phase.
Arm/Group | Enzalutamide | DB Phase: Bicalutamide | Open Label Phase: Bicalutamide Crossover to Enzalutamide
Serious Adverse Events (participants affected / at risk) | 76/197 | 60/198 | 16/37
Other Adverse Events (participants affected / at risk) | 187/197 | 179/198 | 36/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide (N=197) | DB Phase: Bicalutamide (N=198) | Open Label Phase: Bicalutamide Crossover to Enzalutamide (N=37)
Anaemia (Blood and lymphatic system disorders) | 4 | 4 | 2
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 2 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 1 | 1
Angina pectoris (Cardiac disorders) | 5 | 0 | 0
Aortic valve disease (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 5 | 2 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Ileus (Gastrointestinal disorders) | 2 | 0 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 5 | 1 | 0
Chest pain (General disorders) | 2 | 0 | 0
Device occlusion (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 2 | 0
General physical health deterioration (General disorders) | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 3 | 0 | 0
Hepatitis B (Infections and infestations) | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 6 | 4 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 2 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 3 | 1
Septic shock (Infections and infestations) | 1 | 2 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 6 | 1
Urosepsis (Infections and infestations) | 1 | 3 | 0
Fall (Injury, poisoning and procedural complications) | 5 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 1 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 2 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Erythroleukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 0
Cervical cord compression (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 2 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0
Hypoglycaemic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 2 | 0 | 0
Syncope (Nervous system disorders) | 3 | 2 | 1
Transient ischaemic attack (Nervous system disorders) | 5 | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 2 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Bladder obstruction (Renal and urinary disorders) | 0 | 1 | 0
Bladder outlet obstruction (Renal and urinary disorders) | 1 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 5 | 4 | 1
Hydronephrosis (Renal and urinary disorders) | 4 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Postrenal failure (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 2 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0
Vesical fistula (Renal and urinary disorders) | 1 | 0 | 0
Prostatic calcification (Reproductive system and breast disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Accelerated hypertension (Vascular disorders) | 2 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 3 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 2 | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1
Disease progression (General disorders) | 1 | 0 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Urinary bladder abscess (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Urinary bladder rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cystitis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 2
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1
Troponin increased (Investigations) | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 2
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0 | 0
Obstructive uropathy (Renal and urinary disorders) | 1 | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Umbilical hernia repair (Surgical and medical procedures) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide (N=197) | DB Phase: Bicalutamide (N=198) | Open Label Phase: Bicalutamide Crossover to Enzalutamide (N=37)
Abdominal pain (Gastrointestinal disorders) | 15 | 6 | 1
Constipation (Gastrointestinal disorders) | 29 | 33 | 6
Diarrhoea (Gastrointestinal disorders) | 26 | 29 | 9
Nausea (Gastrointestinal disorders) | 38 | 32 | 9
Vomiting (Gastrointestinal disorders) | 12 | 17 | 3
Asthenia (General disorders) | 16 | 5 | 2
Fatigue (General disorders) | 82 | 56 | 10
Pyrexia (General disorders) | 5 | 12 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 45 | 29 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 41 | 34 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 13 | 6 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 16 | 11 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 | 10 | 1
Dizziness (Nervous system disorders) | 26 | 15 | 6
Headache (Nervous system disorders) | 14 | 15 | 1
Anxiety (Psychiatric disorders) | 13 | 3 | 0
Depression (Psychiatric disorders) | 15 | 8 | 2
Insomnia (Psychiatric disorders) | 22 | 9 | 2
Haematuria (Renal and urinary disorders) | 16 | 13 | 3
Renal failure acute (Renal and urinary disorders) | 7 | 12 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 12 | 1
Rash (Skin and subcutaneous tissue disorders) | 12 | 9 | 3
Hot flush (Vascular disorders) | 34 | 20 | 2
Hypertension (Vascular disorders) | 25 | 10 | 5
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 2 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 2 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 22 | 21 | 3
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3 | 0
Branchial cyst (Congenital, familial and genetic disorders) | 1 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 1 | 0 | 0
Type V hyperlipidaemia (Congenital, familial and genetic disorders) | 1 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1
Deafness bilateral (Ear and labyrinth disorders) | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 5 | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1 | 1
Thyroid cyst (Endocrine disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0
Liver injury (Hepatobiliary disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 2 | 1 | 0
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 4 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 4 | 3 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 3 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0
Acquired oesophageal web (Gastrointestinal disorders) | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 1 | 0
Bowel movement irregularity (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0
Defaecation urgency (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 3 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 3 | 2 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 6 | 5 | 1
Dysphagia (Gastrointestinal disorders) | 4 | 4 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 9 | 5 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 4 | 1 | 0
Gastritis (Gastrointestinal disorders) | 8 | 2 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 | 2 | 6
Gingival swelling (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 2 | 0
Hiatus hernia (Gastrointestinal disorders) | 2 | 2 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 2 | 0
Mesenteric artery stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal achalasia (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal dilatation (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal disorder (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 3 | 0 | 0
Pancreatic atrophy (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatic cyst (Gastrointestinal disorders) | 1 | 0 | 0
Rectal discharge (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 1 | 1
Rectal tenesmus (Gastrointestinal disorders) | 0 | 1 | 0
Retching (Gastrointestinal disorders) | 1 | 1 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 1 | 0
Tongue ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Tooth loss (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 3 | 2 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 6 | 2 | 0
Chills (General disorders) | 5 | 2 | 0
Device dislocation (General disorders) | 1 | 0 | 0
Device occlusion (General disorders) | 0 | 1 | 1
Discomfort (General disorders) | 0 | 0 | 1
Early satiety (General disorders) | 3 | 1 | 0
Face oedema (General disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 6 | 1 | 1
Generalised oedema (General disorders) | 0 | 3 | 0
Inflammation (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 5 | 5 | 0
Injection site reaction (General disorders) | 1 | 0 | 0
Local swelling (General disorders) | 4 | 1 | 0
Localised oedema (General disorders) | 2 | 0 | 0
Malaise (General disorders) | 1 | 2 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0
Oedema (General disorders) | 2 | 1 | 0
Oedema peripheral (General disorders) | 17 | 10 | 1
Pain (General disorders) | 7 | 5 | 0
Suprapubic pain (General disorders) | 0 | 0 | 1
Temperature intolerance (General disorders) | 1 | 0 | 0
Thirst (General disorders) | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0
Abscess soft tissue (Infections and infestations) | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 2 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0
Asymptomatic bacteriuria (Infections and infestations) | 1 | 0 | 0
Axillary candidiasis (Infections and infestations) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 1 | 0
Bacterial disease carrier (Infections and infestations) | 0 | 1 | 0
Bacteriuria (Infections and infestations) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 7 | 1 | 0
Candida infection (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 5 | 1 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 3 | 0 | 0
Ear infection (Infections and infestations) | 1 | 2 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 1
Furuncle (Infections and infestations) | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 2 | 0 | 0
Genital infection fungal (Infections and infestations) | 0 | 1 | 0
Gingival infection (Infections and infestations) | 0 | 1 | 0
Gingivitis (Infections and infestations) | 2 | 0 | 0
Helicobacter infection (Infections and infestations) | 1 | 0 | 0
Hepatitis B (Infections and infestations) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 5 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 1 | 0
Incision site infection (Infections and infestations) | 0 | 1 | 0
Infected cyst (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 5 | 1 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0
Mucosal infection (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 8 | 11 | 0
Onychomycosis (Infections and infestations) | 2 | 1 | 0
Oral candidiasis (Infections and infestations) | 2 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 1
Oropharyngitis fungal (Infections and infestations) | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0
Peripheral nerve infection (Infections and infestations) | 1 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 5 | 6 | 1
Postoperative wound infection (Infections and infestations) | 2 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 6 | 5 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0
Tinea infection (Infections and infestations) | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 4 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 8 | 0
Urinary bladder abscess (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 14 | 21 | 7
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contrast media reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 5 | 1 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 1 | 1 | 1
Eschar (Injury, poisoning and procedural complications) | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 3 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 39 | 19 | 8
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 2 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 2 | 0
Laceration (Injury, poisoning and procedural complications) | 10 | 3 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 2 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 4 | 2
Radiation injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 4 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 7 | 6 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 4 | 1 | 0
Splinter (Injury, poisoning and procedural complications) | 1 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vth nerve injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 2 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 5 | 0
Blood albumin decreased (Investigations) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 5 | 11 | 0
Blood bicarbonate decreased (Investigations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 3 | 1 | 0
Blood calcium increased (Investigations) | 0 | 1 | 0
Blood cholesterol increased (Investigations) | 2 | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 6 | 7 | 0
Blood creatinine increased (Investigations) | 5 | 7 | 1
Blood glucose increased (Investigations) | 0 | 3 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 4 | 0
Blood lactic acid increased (Investigations) | 1 | 0 | 0
Blood parathyroid hormone increased (Investigations) | 1 | 0 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0
Blood pressure increased (Investigations) | 3 | 1 | 2
Blood sodium decreased (Investigations) | 1 | 0 | 0
Blood urine present (Investigations) | 1 | 1 | 0
Cardiac murmur (Investigations) | 1 | 1 | 0
Face and mouth X-ray abnormal (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 4 | 1
Helicobacter test positive (Investigations) | 1 | 0 | 0
International normalised ratio fluctuation (Investigations) | 0 | 1 | 0
International normalised ratio increased (Investigations) | 1 | 2 | 0
Intraocular pressure increased (Investigations) | 0 | 1 | 0
Low density lipoprotein increased (Investigations) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 2 | 0 | 0
Lymphocyte count increased (Investigations) | 1 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Neutrophil count increased (Investigations) | 1 | 0 | 0
Occult blood positive (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 4 | 0 | 0
Protein total decreased (Investigations) | 0 | 1 | 0
Protein total increased (Investigations) | 1 | 0 | 0
Red blood cell count decreased (Investigations) | 0 | 1 | 0
Residual urine volume increased (Investigations) | 0 | 1 | 0
Urine ketone body present (Investigations) | 0 | 1 | 0
Urine leukocyte esterase positive (Investigations) | 1 | 1 | 0
Vitamin D increased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 16 | 13 | 3
Weight increased (Investigations) | 1 | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0
White blood cell count increased (Investigations) | 1 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 28 | 17 | 6
Dehydration (Metabolism and nutrition disorders) | 13 | 6 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 2 | 0 | 0
Gout (Metabolism and nutrition disorders) | 3 | 3 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 14 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 4 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 4 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 4 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 13 | 11 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 4 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 10 | 4 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Insulin resistance (Metabolism and nutrition disorders) | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 2 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 2 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 0
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 3 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 2 | 2
Bunion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 6 | 4 | 0
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint crepitation (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 6 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 13 | 4 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 5 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 4 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 | 1 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 4 | 1
Inguinal mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0
Amnesia (Nervous system disorders) | 7 | 0 | 3
Aphasia (Nervous system disorders) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 2 | 0 | 0
Balance disorder (Nervous system disorders) | 3 | 1 | 2
Carotid artery occlusion (Nervous system disorders) | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 1 | 0
Cerebellar infarction (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Cervical radiculopathy (Nervous system disorders) | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 2 | 0 | 1
Dementia (Nervous system disorders) | 2 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 2 | 0 | 0
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 8 | 3 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Essential tremor (Nervous system disorders) | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0
Hypersomnia (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 4 | 3 | 0
Hypogeusia (Nervous system disorders) | 1 | 0 | 0
Hyposmia (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 2 | 0 | 0
Memory impairment (Nervous system disorders) | 8 | 3 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 7 | 0 | 2
Paraesthesia (Nervous system disorders) | 8 | 4 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0 | 0
Parosmia (Nervous system disorders) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0 | 1
Peroneal nerve palsy (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 5 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 2 | 0 | 0
Sciatica (Nervous system disorders) | 3 | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 3 | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0
Visual field defect (Nervous system disorders) | 1 | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 1 | 1 | 0
Muscle spasticity (Nervous system disorders) | 1 | 0 | 0
Periodic limb movement disorder (Nervous system disorders) | 1 | 0 | 0
Post-traumatic headache (Nervous system disorders) | 1 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 2 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0
Alcoholism (Psychiatric disorders) | 0 | 1 | 0
Apathy (Psychiatric disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 6 | 2 | 0
Delirium (Psychiatric disorders) | 1 | 2 | 0
Depressed mood (Psychiatric disorders) | 0 | 2 | 0
Disorientation (Psychiatric disorders) | 0 | 1 | 0
Emotional distress (Psychiatric disorders) | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0
Libido decreased (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 1 | 0
Mood swings (Psychiatric disorders) | 2 | 0 | 0
Nervousness (Psychiatric disorders) | 3 | 0 | 0
Personality change (Psychiatric disorders) | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 3 | 0 | 0
Sleep terror (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0
Bladder neck obstruction (Renal and urinary disorders) | 1 | 0 | 1
Bladder outlet obstruction (Renal and urinary disorders) | 2 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 3 | 0
Calculus bladder (Renal and urinary disorders) | 2 | 1 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 2 | 7 | 0
Enuresis (Renal and urinary disorders) | 0 | 1 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 6 | 8 | 1
Hypertonic bladder (Renal and urinary disorders) | 1 | 0 | 0
Incontinence (Renal and urinary disorders) | 2 | 0 | 0
Microalbuminuria (Renal and urinary disorders) | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 9 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 3 | 1 | 0
Nocturia (Renal and urinary disorders) | 3 | 4 | 2
Oliguria (Renal and urinary disorders) | 0 | 1 | 0
Pneumaturia (Renal and urinary disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 11 | 7 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Pyuria (Renal and urinary disorders) | 0 | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 3 | 0
Renal failure chronic (Renal and urinary disorders) | 3 | 1 | 1
Renal impairment (Renal and urinary disorders) | 0 | 2 | 0
Renal pain (Renal and urinary disorders) | 1 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 1 | 1 | 0
Urethral haemorrhage (Renal and urinary disorders) | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 2 | 0
Urethritis noninfective (Renal and urinary disorders) | 0 | 1 | 0
Urge incontinence (Renal and urinary disorders) | 1 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 10 | 8 | 1
Urinary retention (Renal and urinary disorders) | 5 | 7 | 0
Urinary tract obstruction (Renal and urinary disorders) | 3 | 3 | 0
Urine flow decreased (Renal and urinary disorders) | 1 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 1 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0
Genital discomfort (Reproductive system and breast disorders) | 1 | 0 | 0
Genital lesion (Reproductive system and breast disorders) | 1 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 2 | 2 | 0
Nipple pain (Reproductive system and breast disorders) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 1 | 0
Penile oedema (Reproductive system and breast disorders) | 1 | 0 | 0
Penile swelling (Reproductive system and breast disorders) | 0 | 1 | 0
Priapism (Reproductive system and breast disorders) | 1 | 0 | 0
Prostatic pain (Reproductive system and breast disorders) | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 0
Scrotal swelling (Reproductive system and breast disorders) | 0 | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 4 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Alveolar lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 9 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pulmonary vascular disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 3 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 2 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 3 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 | 2 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Lentigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Photodermatosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 3 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Cataract operation (Surgical and medical procedures) | 1 | 0 | 0
Skin neoplasm excision (Surgical and medical procedures) | 0 | 1 | 1
Accelerated hypertension (Vascular disorders) | 1 | 1 | 0
Aortic arteriosclerosis (Vascular disorders) | 1 | 0 | 0
Arteriovenous fistula (Vascular disorders) | 1 | 0 | 0
Blood pressure inadequately controlled (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 1 | 1
Flushing (Vascular disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 1 | 1 | 1
Hypotension (Vascular disorders) | 4 | 5 | 4
Intermittent claudication (Vascular disorders) | 1 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 2 | 2 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 1 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 2 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 1
Bone contusion (Injury, poisoning and procedural complications) | 3 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 1 | 0
Blood urea increased (Investigations) | 1 | 2 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 1
Syncope (Nervous system disorders) | 7 | 3 | 1
Angina pectoris (Cardiac disorders) | 2 | 1 | 0
Aortic valve disease (Cardiac disorders) | 1 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 5 | 3
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Atrial thrombosis (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 2 | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 4 | 3 | 2
Cardiomegaly (Cardiac disorders) | 0 | 1 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 2 | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 3 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Astigmatism (Eye disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 4 | 3 | 1
Cataract nuclear (Eye disorders) | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 3 | 0 | 1
Diabetic retinopathy (Eye disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 1
Eye irritation (Eye disorders) | 1 | 1 | 0
Eye pain (Eye disorders) | 1 | 0 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 3 | 0 | 0
Macular degeneration (Eye disorders) | 1 | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 1 | 0
Photophobia (Eye disorders) | 1 | 0 | 0
Posterior capsule opacification (Eye disorders) | 0 | 1 | 0
Retinal tear (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 4 | 2 | 0
Visual impairment (Eye disorders) | 4 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees not to independently publish the results before the publication of the multi-center PI paper. Sponsor shall review and comment 30 days prior to submission or disclosure. If publication or disclosure contains Sponsor Confidential Information, other than study data, PI agrees to remove Confidential Information from publication or disclosure. Sponsor may request that PI delay such publication for an additional 60 days to protect the patentability of any invention described.